CLINICAL TRIAL: NCT01414192
Title: Model-Observation Bridging Study (MOBS) for Ezetrol® and Inegy®
Brief Title: A Study to Design a Model Cohort for Analysis of Dyslipidemia (MK-0653A-204)
Acronym: MOBS
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0653A-204
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2022-02

CONDITIONS: Dyslipidemia; Hypercholesterolemia
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Ezetimibe monotherapy without prior treatment: Enrolled participants who had no prior lipid-lowering therapy and were currently receiving Ezetimibe alone (Ezetrol®).
- Ezetimibe monotherpay with prior treatment: Enrolled participants with prior lipid-lowering therapy and were currently receiving Ezetimibe alone (Ezetrol®).
- Ezetimibe plus statin: Enrolled participants who were being coadministered ezetimide (Ezetrol®) and another prescription statin.
- Ezetimibe/simvastatin: Enrolled participants who were receiving ezetimibe and simavastatin fixed dose combination tablet (Inegy®).

SUMMARY:
This study is being done to provide valid data on the evolution of a cohort of French participants treated with ezetimibe, alone or in combination with a statin, to be used in simulation models for cardiovascular disease (CVD). Patterns of drug use, evolution of risk factors for CVD, cardiovascular morbidity and mortality, and goal attainment in low density lipoprotein cholesterol (LDL-C) levels over time will be analyzed.

ELIGIBILITY:
Inclusion criteria:

* Resident of Continental France
* Treated by ezetimibe either as monotherapy (Ezetrol®), or co-administered with a statin or administered in a fixed combination of ezetimibe and simvastatin (Inegy®)
* Incident treatment with ezetimibe at the time of recruitment into the study

Exclusion criteria:

* Unlikely to be followed-up for the next 6 months after recruitment due to a planned change of residence
* Participating in a clinical trial
* Unable to read the information letter in French and/or unable to participate in the telephone interview in French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The resident population of Continental France being treated for hypercholesterolemia in a general practice setting.
Sampling Method: Non-Probability Sample
Enrollment: 3215 (Actual)
Dates: Start 2008-11-15 (Actual); Primary Completion 2014-09-15 (Actual); Study Completion 2014-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Ferrieres J, Dallongeville J, Rossignol M, Benichou J, Caro JJ, Getsios D, Hernandez L, Abenhaim L, Grimaldi-Bensouda L. Model-observational bridging study on the effectiveness of ezetimibe on cardiovascular morbidity and mortality in France: A population-based study. J Clin Lipidol. 2016 Nov-Dec;10(6):1379-1388. doi: 10.1016/j.jacl.2016.08.015. Epub 2016 Sep 7. PMID 27919355

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data was provided by French physicians for participants who were being administered Ezetrol® monotherapy, or Ezetrol® coadministered with a statin, or Inegy® (a fixed-dose combination of ezetimibe and simvastatin.
Pre-assignment Details: All participants who met inclusion criteria and contributed to at least one type of follow-up data in the form of an interview or physician questionnaire were included in the study.
Groups:
- Ezetimibe Plus Statin: Enrolled participants who were being coadministered ezetimide (Ezetrol®) and another prescription statin or ezetimide with simvastatin
Period: Overall Study
Arm/Group | Ezetimibe Monotherapy Without Prior Treatment | Ezetimibe Monotherpay With Prior Treatment | Ezetimibe Plus Statin | Ezetimibe/Simvastatin
Started | 490 | 575 | 424 | 1726
Completed | 490 | 575 | 424 | 1726
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe Monotherapy Without Prior Treatment | Ezetimibe Monotherpay With Prior Treatment | Ezetimibe Plus Statin | Ezetimibe/Simvastatin | Total
Number analyzed (Participants) | 490 | 575 | 424 | 1726 | 3215
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (11.5) | 63.3 (9.7) | 60.8 (10.8) | 61.4 (10.6) | 61.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 283 | 284 | 164 | 728 | 1459
  Male | 207 | 291 | 260 | 998 | 1756

OUTCOME MEASURES:

1. Primary Outcome: Rate of Cardiovascular (CV) Events
Description: Number of participants who experienced myocardial infarction, acute coronary syndrome, unstable angina, ischemic stroke, revascularization procedure, fatal stroke, and/or sudden death was recorded. The number of events was divided by the total number of patient-years calculated for each treatment group to produce the rate of CV events per 1000 patient years.
Time Frame: up to 48 months
Population: All participants with available data for endpoint.
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Groups:
- Ezetimibe Monotherapy With Prior Treatment: Enrolled participants who had prior lipid-lowering therapy and were currently receiving Ezetimibe alone (Ezetrol®).
Arm/Group | Ezetimibe Monotherapy Without Prior Treatment | Ezetimibe Monotherapy With Prior Treatment | Ezetimibe Plus Statin | Ezetimibe/Simvastatin
Number analyzed (Participants) | 490 | 575 | 424 | 1726
Events per 1000 patient-years | 7.91 [3.95 to 14.14] | 10.79 [6.39 to 17.05] | 12.77 [7.3 to 20.74] | 13.4 [10.38 to 17.01]

2. Secondary Outcome: Percentage Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) Levels at 12 Months
Description: LDL-C levels at baseline and after 12 months of treatment were compared and the percentage change was recorded. In the model, it is assumed that the 5th and 95th percentiles represent the minimum and maximum effect of treatment, respectively.
Time Frame: Baseline and Month 12
Population: All participants with available data for endpoint. The ezetimibe plus statin and ezetimibe/simvastatin arms were combined for this outcome.
Measure: Mean (Full Range); unit: Percentage Change
Groups:
- Ezetimibe Plus Statin or Ezetimibe/Simvastatin: Enrolled participants who were being coadministered ezetimide (Ezetrol®) and another prescription statin or ezetimide with simvastatin or were receiving ezetimibe and simavastatin fixed dose combination tablet (Inegy®).
Arm/Group | Ezetimibe Monotherapy Without Prior Treatment | Ezetimibe Monotherapy With Prior Treatment | Ezetimibe Plus Statin or Ezetimibe/Simvastatin
Number analyzed (Participants) | 490 | 575 | 2150
Percentage Change | -22.4 [-51.6 to 8.2] | -7.1 [-45.6 to 47.0] | -30.7 [-63.6 to 16.1]

3. Secondary Outcome: Percentage of Participants With CV Risk Factors
Description: Enrolled participants' data were reviewed for presence of CV risk factors that included smoking, alcohol & substance abuse, high blood pressure, Type 1 and Type 2 diabetes mellitus, cholesterol level, hypertriglyceridemia, body mass index, cardiovascular disease history, family history of early cardiovascular disease. The sum of all risk factors was tabulated for each participant and totals were summarized by group.
Time Frame: At enrollment (baseline)
Population: All enrolled participants with available data
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe Monotherapy Without Prior Treatment | Ezetimibe Monotherapy With Prior Treatment | Ezetimibe Plus Statin | Ezetimibe/Simvastatin
Number analyzed (Participants) | 490 | 575 | 424 | 1726
Percentage of Participants
  0 risk factors | 19.0 | 15.0 | 11.3 | 11.2
  1 risk factor | 29.0 | 20.9 | 19.6 | 21.8
  2 risk factors | 30.6 | 34.1 | 32.5 | 31.9
  3 risk factors | 16.3 | 22.1 | 25.9 | 23.6
  4 risk factors | 4.3 | 7.0 | 8.3 | 9.2
  5 risk factors | 0.8 | 1.0 | 2.4 | 2.2
  6 risk factors | 0.0 | 0.0 | 0.0 | 0.1

4. Secondary Outcome: Percentage of Participants Who Continued Treatment for 12, 24, 36, and 48 Months
Description: Participants' data reviewed and the number of participants who had continued treatment for 12, 24, 36, and 48 months was recorded.
Time Frame: up to 48 months
Population: All enrolled participants with available data. The ezetimibe monotherapy with or without previous lipid-lowering treatment groups were combined for this outcome.
Measure: Number; unit: Percentage of Participants
Groups:
- Ezetimibe Monotherapy With or Without Prior Treatment: Enrolled participants with or without prior lipid-lowering therapy and were currently receiving Ezetimibe alone (Ezetrol®).
Arm/Group | Ezetimibe Monotherapy With or Without Prior Treatment | Ezetimibe Plus Statin | Ezetimibe/Simvastatin
Number analyzed (Participants) | 1065 | 424 | 1726
Percentage of Participants
  12 months (n=857; 446; 1755) | 28.0 | 14.6 | 57.4
  24 months (n=722; 380; 1563) | 27.1 | 14.3 | 58.6
  36 months (n=433; 248; 1025) | 25.4 | 14.5 | 60.1
  48 months (n=203; 127; 437) | 26.5 | 16.6 | 57.0

5. Secondary Outcome: Percentage of Participants With at Least 1 Discontinuation of Study Drug
Description: The percentage of participants who stopped study drug at least once during the study period was recorded and summarized.
Time Frame: up to 48 months
Population: All enrolled participants with available data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ezetimibe Monotherapy Without Prior Treatment | Ezetimibe Monotherapy With Prior Treatment | Ezetimibe Plus Statin | Ezetimibe/Simvastatin
Number analyzed (Participants) | 490 | 575 | 424 | 1726
Percentage of Participants | 15.8 | 13.4 | 10.1 | 11.8

6. Secondary Outcome: Mortality Rate
Description: The number of participants who died from any cause was recorded. The number of deaths was then extrapolated to produce the number of deaths per 100,000 patient-years.
Time Frame: up to 48 months
Population: All enrolled participants with available data.
Measure: Number (95% Confidence Interval); unit: Deaths per 100,000 patient-years
Arm/Group | Ezetimibe Monotherapy Without Prior Treatment | Ezetimibe Monotherapy With Prior Treatment | Ezetimibe Plus Statin | Ezetimibe/Simvastatin
Number analyzed (Participants) | 378 | 452 | 342 | 1369
Deaths per 100,000 patient-years | 506.54 [185.89 to 1102.53] | 689.66 [330.72 to 1268.30] | 817.81 [373.95 to 1552.46] | 761.77 [524.37 to 1069.81]

ADVERSE EVENTS:
Description: There was no plan to systematically collect adverse events for this study.
Arm/Group | Ezetimibe Monotherapy Without Prior Treatment | Ezetimibe Monotherapy With Prior Treatment | Ezetimibe Plus Statin | Ezetimibe/Simvastatin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No